CLINICAL TRIAL: NCT00174967
Title: Phase II, Dose-Response, Safety and Efficacy Study of Oral TMX-67 in Subjects With Gout.
Brief Title: Dose-Response, Safety and Efficacy of Febuxostat in Subjects With Gout
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: TMX-00-004; U1111-1114-1992 (Registry Identifier: WHO)
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2009-07-16 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Gout
Keywords: Uric Acid; xanthine oxidase; tophi; Drug Therapy
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo
- Febuxostat 40 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Febuxostat 80 mg QD (Experimental)
  Interventions: Drug: Febuxostat
- Febuxostat 120 mg QD (Experimental)
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Placebo — Febuxostat placebo-matching tablets, orally, once daily for up to 4 weeks.
  Arms: Placebo QD
Drug: Febuxostat — Febuxostat 40 mg, tablets, orally, once daily for up to 4 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 40 mg QD
Drug: Febuxostat — Febuxostat 80 mg, tablets, orally, once daily for up to 4 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 80 mg QD
Drug: Febuxostat — Febuxostat 120 mg, tablets, orally, once daily for up to 4 weeks.
  Other Names: TMX-67; Tei-6720; Uloric
  Arms: Febuxostat 120 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy of febuxostat, once daily (QD), in reducing serum urate levels in subjects with gout.

DETAILED DESCRIPTION:
Gout is a chronic urate crystal deposition disorder, which if left untreated may result in progressive disease characterized by joint and bone destruction from tophaceous deposits and renal impairment due to gouty nephropathy. Hyperuricemia, defined as a serum urate concentration of >7.0 milligrams per deciliter (mg/dL), is the underlying metabolic aberration leading to urate crystal deposition in gout. Gout has several clinical presentations, including: recurrent acute attacks of inflammatory arthritis; deposition of monosodium urate monohydrate crystals in joints, bones and even parenchymal organs (tophaceous gout); renal impairment; and uric acid nephrolithiasis. As serum urate levels increase beyond >7.0 mg/dL, the risks for gouty arthritis or for renal calculi increase.

Currently allopurinol is the only xanthine oxidase inhibitor available. Allopurinol is the agent of choice for reduction of serum urate levels in patients with: uric acid overproduction; unresponsive or intolerant to uricosuric agents; impaired renal function; uric acid urolithiasis; or tophi.

Febuxostat (TMX-67) is a non-purine selective xanthine oxidase inhibitor being developed as an orally administered agent for management of hyperuricemia in patients with gout.

ELIGIBILITY:
Inclusion Criteria:

* Hyperuricemia (serum uric acid ≥8.0 mg/dL).
* Must meet American College of Rheumatology criteria for gout.
* Must have adequate renal function (serum creatinine <1.5 mg/dL).
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* History of xanthinuria
* Alcohol consumption >14/week
* Has a history of significant concomitant illness.
* Has active liver disease.
* Has a body mass index greater than 50 kilogram per meter² (kg/m²)
* Any other significant medical condition that would interfere with the treatment, safety or compliance with the protocol, as defined by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2001-01; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Takeda

REFERENCES:
- [Result] Becker MA, Schumacher HR Jr, Wortmann RL, MacDonald PA, Palo WA, Eustace D, Vernillet L, Joseph-Ridge N. Febuxostat, a novel nonpurine selective inhibitor of xanthine oxidase: a twenty-eight-day, multicenter, phase II, randomized, double-blind, placebo-controlled, dose-response clinical trial examining safety and efficacy in patients with gout. Arthritis Rheum. 2005 Mar;52(3):916-23. doi: 10.1002/art.20935. PMID 15751090
- [Result] Colwell HH, Hunt BJ, Pasta DJ, Palo WA, Mathias SD, Joseph-Ridge N. Gout Assessment Questionnaire: Initial results of reliability, validity and responsiveness. Int J Clin Pract. 2006 Oct;60(10):1210-7. doi: 10.1111/j.1742-1241.2006.01104.x. Epub 2006 Aug 15. PMID 16911575
- [Result] Goldfarb DS, MacDonald PA, Hunt B, Gunawardhana L. Febuxostat in gout: serum urate response in uric acid overproducers and underexcretors. J Rheumatol. 2011 Jul;38(7):1385-9. doi: 10.3899/jrheum.101156. Epub 2011 May 15. PMID 21572152
- See also: Uloric Package Insert — http://general.takedapharm.com/content/file.aspx?applicationcode=6C7C39D8-5D09-453B-BF30-696A4AB88E62&fileTypeCode=ULORICPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 24 investigative sites from 31 January 2001 to 9 July 2001
Pre-assignment Details: Participants currently receiving urate-lowering therapy discontinued those urate-lowering therapies and initiated prophylactic medications before enrollemnt in once daily (QD) treatment groups. All other subjects also initiated prophylactic medications.
Groups:
- Febuxostat 40 mg QD: Febuxostat 40 mg, orally, once daily.
- Febuxostat 80 mg QD: Febuxostat 80 mg, orally, once daily.
- Febuxostat 120 mg QD: Febuxostat 120 mg, orally, once daily.
- Placebo QD: Placebo, orally, once daily
Period: Overall Study
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Started | 37 | 40 | 38 | 38
Completed | 36 | 37 | 36 | 36
Not Completed | 1 | 3 | 2 | 2
Not completed — Adverse Event | 1 | 2 | 2 | 1
Not completed — Gout Flare | 0 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD | Total
Number analyzed (Participants) | 37 | 40 | 38 | 38 | 153
Age Continuous [Mean (Standard Deviation); unit: years] | 52.2 (14.04) | 55.2 (13.09) | 56.2 (10.83) | 52.4 (12.63) | 54.0 (12.69)
Age, Customized [Number; unit: participants]
  <45 years | 8 | 10 | 7 | 12 | 37
  45 years to <65 years | 21 | 19 | 23 | 17 | 80
  ≥65 years | 8 | 11 | 8 | 9 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 6 | 17
  Male | 33 | 38 | 33 | 32 | 136
Race/Ethnicity, Customized [Number; unit: participants]
  White | 32 | 35 | 34 | 32 | 133
  Black or African American | 3 | 3 | 2 | 3 | 11
  Hispanic | 1 | 1 | 1 | 1 | 4
  Asian | 0 | 1 | 1 | 0 | 2
  Other | 1 | 0 | 0 | 2 | 3
Body Mass Index [Number; unit: participants]
  ≤25 kilogram per meter² (kg/m²) | 2 | 3 | 3 | 0 | 8
  >25 kg/m² to 30 kg/m² | 12 | 12 | 14 | 13 | 51
  >30 kg/m² to 35 kg/m² | 16 | 12 | 12 | 16 | 56
  >35 kg/m² to 40 kg/m² | 4 | 7 | 5 | 6 | 22
  >40 kg/m² | 3 | 6 | 3 | 3 | 15
  missing | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Whose Serum Urate Level Decreased to <6.0 Milligram Per Deciliter (mg/dL) at the Day 28 Visit.
Description: Serum urate values were obtained at the Day 28 visit. The percentage of subjects whose serum urate decreased to <6.0 mg/dL at the Day 28 visit was summarized.
Time Frame: Day 28.
Population: Analysis performed on intent-to-treat (ITT) subjects, defined as all randomized subjects who took at least 1 dose of study drug and who had baseline serum urate ≥8.0 mg/dL. The last observation carried forward (LOCF) method was used to impute missing data. The baseline value was carried forward if no postbaseline visits were available.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percentage of subjects | 56 | 76 | 94 | 0
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — Pairwise comparisons between placebo and each of the febuxostat treatment groups were performed using Fisher's exact test. Adjustment for multiple comparisons was made using Hochberg's procedure
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Subjects Whose Serum Urate Level Decreased to <6.0 mg/dL at the Day 7 Visit.
Description: Serum urate values were obtained at the Day 7 visit. The percentage of subjects whose serum urate decreased to <6.0 mg/dL at the Day 7 visit was summarized.
Time Frame: Day 7.
Population: The analysis was performed on ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had baseline serum urate ≥ 8.0 mg/dL. The LOCF method was used to impute missing data. The baseline value was carried forward if no post-baseline visits were available.
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percentage of subjects | 50 | 59 | 91 | 3
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Subjects Whose Serum Urate Level Decreased to <6.0 mg/dL at the Day 14 Visit.
Description: Serum urate values were obtained at the Day 14 visit. The percentage of subjects whose serum urate decreased to <6.0 mg/dL at the Day 14 visit was summarized.
Time Frame: Day 14.
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percentage of subjects | 56 | 68 | 94 | 0
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Subjects Whose Serum Urate Level Decreased to <6.0 mg/dL at the Day 21 Visit.
Description: Serum urate values were obtained at the Day 21 visit. The percentage of subjects whose serum urate decreased to <6.0 mg/dL at the Day 21 visit was summarized.
Time Frame: Day 21.
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percentage of subjects | 59 | 76 | 97 | 0
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Fisher Exact — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline to the Day 7 Visit.
Description: Serum urate values were obtained at the Day 7 visit. The percent change in serum urate from baseline to the Day 7 visit was summarized.
Time Frame: Baseline and Day 7.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percent change from baseline | -35.0 (9.67) | -39.2 (15.9) | -53.44 (12.3) | 0.71 (12.6)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Pairwise comparisons between placebo and each of the febuxostat treatment groups were performed using a t-test. Adjustment for multiple comparisons was made using Hochberg's procedure
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline to the Day 14 Visit.
Description: Serum urate values were obtained at the Day 14 visit. The percent change in serum urate from baseline to the Day 14 visit was summarized.
Time Frame: Baseline and Day 14.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percent change from baseline | -37.1 (11.70) | -41.8 (14.63) | -56.9 (8.36) | 1.62 (10.21)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline to the Day 21 Visit
Description: Serum urate values were obtained at the Day 21 visit. The percent change in serum urate from baseline to the Day 21 visit was summarized.
Time Frame: Baseline and Day 21.
Population: The analysis was performed on ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had baseline serum urate ≥ 8.0 mg/dL. The last observation carried forward (LOCF) method was used to impute missing data. The baseline value was carried forward if no post-baseline visits were available.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percent change from baseline | -37.3 (11.30) | -43.9 (16.3) | -59.4 (7.58) | -0.57 (10.63)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]

8. Secondary Outcome: Percent Change in Serum Urate Levels From Baseline to the Day 28 Visit.
Description: Serum urate values were obtained at the Day 28 visit. The percent change in serum urate from baseline to the Day 28 visit was summarized.
Time Frame: Baseline and Day 28.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percent change from baseline | -36.6 (12.07) | -44.3 (17.53) | -59.1 (9.92) | -2.2 (12.5)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]

9. Secondary Outcome: Maximum Percent Change in Serum Urate Level From Baseline During the Entire Treatment Period.
Description: Serum urate values were obtained at the Day 7, 14, 21,and 28 visits. The maximum percent change in serum urate levels obtained at any visit was summarized.
Time Frame: Baseline and Any visit (Day 7, 14, 21,or 28)
Population: The analysis was performed on ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had baseline serum urate ≥ 8.0 mg/dL.
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 34 | 37 | 34 | 35
percent change from baseline | 42.5 (10.04) | 49.2 (13.24) | 62.8 (7.05) | 10.0 (11.12)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]

10. Secondary Outcome: Percent Change in 24-hour Urine Uric Acid Level From Baseline to Day 28.
Description: 24-hour urine uric acid levels were obtained at the Day 28 visit. The percent change in 24-hour urine uric acid level from baseline to the Day 28 visit was summarized.
Time Frame: Baseline and Day 28.
Population: The analysis was performed on ITT subjects, which were defined as all randomized subjects who took at least 1 dose of study drug and who had baseline serum urate ≥ 8.0 mg/dL. Missing data was not imputed
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Number analyzed (Participants) | 33 | 35 | 34 | 34
percent change from baseline | -43.6 (28.9) | -46.5 (27.0) | -45.7 (30.1) | 5.9 (37.1)
Statistical Analysis 1: Comparison: Febuxostat 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Febuxostat 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Febuxostat 120 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Arm/Group | Febuxostat 40 mg QD | Febuxostat 80 mg QD | Febuxostat 120 mg QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/40 | 2/38 | 0/38
Other Adverse Events (participants affected / at risk) | 18/37 | 19/40 | 16/38 | 17/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 40 mg QD (N=37) | Febuxostat 80 mg QD (N=40) | Febuxostat 120 mg QD (N=38) | Placebo QD (N=38)
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Delirium (Nervous system disorders) | 0 | 1 | 0 | 0
Guillian Barre Syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Back Pain (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Febuxostat 40 mg QD (N=37) | Febuxostat 80 mg QD (N=40) | Febuxostat 120 mg QD (N=38) | Placebo QD (N=38)
Abdominal Pain (General disorders) | 1 | 1 | 2 | 3
Accidental Injury (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Back Pain (General disorders) | 3 | 2 | 2 | 1
Flu Syndrome (General disorders) | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 3 | 2 | 2 | 1
Infection (Infections and infestations) | 1 | 0 | 1 | 2
Pain (General disorders) | 6 | 3 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 4 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Increased Appetite (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Liver Function Tests Abnormal (Investigations) | 2 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.